CLINICAL TRIAL: NCT01799876
Title: Autologous Cell Therapy Enhancement of Microfracture Surgery
Brief Title: Use of Cell Therapy to Enhance Arthroscopic Knee Cartilage Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondren Orthopedic Group L.L.P. (Other)
Collaborators: InGeneron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOG-TOH125
Record Dates: First submitted 2013-02-22; First posted 2013-02-27 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Articular Cartilage Defect Grade III or IV of the Knee
Keywords: knee; cartilage; microfracture; cell therapy
MeSH Terms: conditions — Fractures, Stress | interventions — FANG vaccine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Cell (Experimental): Regenerative cells obtained from autologous fat are administered in the knee at microfracture site.
  Interventions: Procedure: Autologous Cell
- Control (Sham Comparator): Standard arthroscopy with sham lipoplasty procedure (no fat cells harvested).
  Interventions: Procedure: Standard microfracture arthroscopic surgery

INTERVENTIONS:
Procedure: Autologous Cell
  Arms: Autologous Cell
Procedure: Standard microfracture arthroscopic surgery
  Arms: Control

SUMMARY:
The purpose of this study is to assess the potential benefit of enhancing knee surgery for cartilage injury using some of the patient's own cells, taken from fat tissue, that may be able to help cartilage to regenerate.

DETAILED DESCRIPTION:
Participation in this study will allow the surgical team to remove a small amount of fat (20 to 30 ml, or between 1 and 2 tablespoons) from just below the skin in the belly region that will be processed to remove regenerative cells, which will then inserted into the knee to the damaged cartilage. These cells may encourage healing at the surgical site, although whether or how much they encourage healing is unknown. Determining whether such improved healing occurs is the purpose of this study.

Some patients will have the fat removed and cells inserted in their knee, and other patients will not have the fat removed or cells inserted. To which group patients are assigned is determined by a random process, similar to flipping a coin. The surgery is the same in all other ways for all patients.

Participation will require attending regularly scheduled postoperative visits, having 3 MRI tests, and answering a short survey. No additional visits other beyond those normally scheduled for postsurgical care are required.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing microfracture surgery for the repair of articular cartilage
* Osteochondral defect Grade III or IV
* Age 18 to 68 years
* Sufficient subcutaneous adipose tissue to yield 20-30 cc of lipoaspirate
* Written informed consent
* Ability to speak, read and write English or Spanish

Exclusion Criteria:

* Inability to speak, read and write English or Spanish
* Evidence of malignant disorder/neoplasm in past 24 months
* History of basal cell carcinoma
* History of smoking and not committed to give up
* Chronic skin conditions
* Connective, metabolic or skin disease
* Evidence of active infection
* Pregnancy or lactating for female subjects
* Diabetes Type I or II
* Current steroid use
* Immunosuppressive medication
* Renal failure (creatine > 1.8 mg/dL)
* Hepatic failure (AST, ALT >2 times normal values; bilirubin >2.0 mg/dL)
* Inflammatory joint diseases of the knee that indicate additional, conflating therapies
* Joint infection within the past 6 months
* Meniscal resection of greater than 50% prior to, or at time of procedure
* Uncorrected joint instability
* Joint malalignment > 5 degrees

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) for osteochondral defect filling | 12 months
  Filling will be scored by quartile with 1 point for less than 25% filling of the defect and 4 points for greater than 75% filling. Evaluated by radiologist who is blinded to group assignment.

SECONDARY OUTCOMES:
Pain Scores on Numerical Rating Scale | up to 1 year
Knee Injury and Osteoarthritis Outcomes Survey (KOOS) | 12 months postop
  Survey
Knee Range of Motion | up to 1 year
Number of Patients with Adverse Events as a Measure of Safety | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Burke, MD, Principal Investigator — Fondren Orthopedic Group L.L.P.
Locations (1):
- Fondren Orthopedic Group, L.L.P., Houston, Texas, United States